CLINICAL TRIAL: NCT00296101
Title: Interventions to Increase Adolescent Physical Activity
Brief Title: School-Based Intervention to Increase Physical Activity Among Adolescent Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 359; R01HL063861-05 (NIH)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2006-02

CONDITIONS: Cardiovascular Diseases; Obesity
Keywords: Physical Inactivity
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Sedentary Behavior | interventions — Exercise

INTERVENTIONS:
Behavioral: Physical Activity

SUMMARY:
Physical inactivity is a major public health problem in the United States. Research has shown that physical activity levels decline during adolescence, and the decline is greater in females than males. The purpose of this study is to evaluate a life-skills oriented physical activity intervention at increasing activity levels and decreasing cardiovascular risk factors in adolescent females.

DETAILED DESCRIPTION:
Physical activity levels decline dramatically during adolescence, particularly among females, with the decline most apparent among African Americans. The health benefits of regular physical activity are well-known; individuals who are active have lower rates of obesity and less incidence of cardiovascular disease. Because physical activity behaviors often develop during childhood, it is important to develop programs specifically for adolescents to encourage them to adopt and maintain a physically active lifestyle. Unfortunately, few programs have been developed that specifically focus on adolescents, and the long-term effectiveness of these programs is unknown. This study will evaluate the effectiveness of a life-skills oriented Comprehensive Physical Activity Program (CAP) at increasing activity levels in adolescents. Participants in the CAP program will develop new behavioral skills, which will assist them to continue a physically active lifestyle once the program ends. The purpose of this study is to compare CAP versus a standard physical education (PE) class at increasing physical activity levels and decreasing cardiovascular risk factors in adolescent African American and Caucasian females.

This study will enroll 9th grade female students who attend a high school in Baltimore, Maryland. They will be randomly assigned to participate in either a standard PE class or CAP. Participants in the CAP program will also receive support from a family member to ensure that they receive encouragement for engaging in exercise. Baseline assessments will include physical activity level; cardiorespiratory fitness; cardiovascular risk factors, including blood pressure, lipoproteins, and body mass index (BMI); and psychosocial factors. Participants will attend follow-up visits at the end of each school year in the 9th, 10th, and 11th grades.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in 9th grade at the participating high school in Baltimore, Maryland

Exclusion Criteria:

* Has a chronic medical disorder
* Currently taking medications that affect the cardiovascular or metabolic systems (e.g., beta adrenergic blockers)
* Excused from the State of Maryland's PE requirement
* Planning on leaving the area prior to the end of the study
* Has a sibling enrolled in the study
* Pregnant or breast-feeding

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300
Dates: Start 2000-02; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Physical activity
Cardiorespiratory fitness (measured at follow-up evaluation 2 1/2 years after study entry)

SECONDARY OUTCOMES:
Sedentary behaviors
Cardiovascular risk factors (measured by blood pressure, lipoproteins, and BMI)
Psychosocial factors (measured at follow-up evaluation 2 1/2 years after study entry)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah R. Young, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, College Park, Maryland, United States